CLINICAL TRIAL: NCT04845126
Title: Outcomes of Patients With Heart Failure Hospitalized in an Internal Medicine Unit - a Four Years Follow-up Study
Brief Title: Outcomes of Patients With Heart Failure Hospitalized in an Internal Medicine Unit
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0188
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure
Keywords: Outcomes; Internal medecine; Heart failure treatment; Heart failure guidelines; quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2018, the investigators evaluated the treatment of 236 patients with heart failure (with preserved or reduced ejection fraction) before and after hospitalization in our internal medicine unit (from 2016 to 2017).

The investigators showed that patients, mainly elderly women with comorbidities, often had suboptimal heart failure treatment without an identified cause. The investigators tried, whenever possible, to optimize treatment before hospital discharge.

Our objective is now to analyze the 4-year outcome of these patients, including re-hospitalization for heart failure or death.

ELIGIBILITY:
Inclusion criteria:

- Patients hospitalized in our Internal Medecine unit for acute heart failure or for another cause but with known chronic heart Failure

Exclusion criteria:

- Hemodilaysis, end stage kidney disease, heart failure cause by anuria, heart transplantation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for heart failure or with known heart failure in our Internal Medecine unit between 2016/01/01 and 2018/01/01.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
re-hospitalization for heart failure or death failure assessed by spirometry | 1 day
  re-hospitalization for heart failure or death (yes or no) (composite outcome)

SECONDARY OUTCOMES:
time to re-hospitalization | 1 day
  time to re-hospitalization
time to death | 1 day
  time to death
cause of hospitalization | 1 day
  cause of hospitalization
cause of death | 1 day
  cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fesler, PUPH, Study Director — UH MONTPELLIER
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC